CLINICAL TRIAL: NCT06639932
Title: Evaluating the Effects of the We-INtervention Among Chinese HIV-serodiscordant Male Couples in a Randomized Controlled Trial
Brief Title: We-INtervention Among Chinese HIV-serodiscordant Male Couples
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: City University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Nancy Xiaonan Yu, Professor, City University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: We-INtervention
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: HIV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- We-INtervention group (Experimental): The interventionists at each study site will be either healthcare providers (e.g., nurses), social workers, or psychologists with at least 3 years of experience serving HIV-serodiscordant male couples.
  Interventions: Behavioral: We-INtervention
- Usual care group (Active Comparator): The participants in the control condition will receive regular care.
  Interventions: Behavioral: Usual Care Group

INTERVENTIONS:
Behavioral: We-INtervention — The We-INtervention focuses on the relationship dynamics of HIV-serodiscordant male couples. In developing the intervention, we reviewed relevant theories and frameworks, such as the cognitive transactional model, the systemic transactional model, the dyadic illness management model, and the intersectional framework of stigma. The three weekly 60-minute sessions are Session 1: We-disease appraisal. Despite stigma related to their dual minority identities, couples develop a perception of HIV as a shared disease, enhancing illness control. Session 2: Couple communication. Couples undertake skill-building exercises on effective communication techniques to strengthen their relationship. Session 3: Dyadic coping. Couples learn to optimize preference and value assessments in HIV management. A few skill-building exercises help them mobilize and maintain mutual support and develop joint problem-solving skills.
  Arms: We-INtervention group
Behavioral: Usual Care Group — The participants in the control condition will receive health information pamphlets. The HIV-seropositive partners will receive information on HIV-related knowledge (e.g., symptoms, comorbidity, stages, and opportunistic infection), treatment (e.g., ART and side effects), and management (e.g., nutrition and mental health). The HIV-seronegative partner will receive information on HIV transmission (e.g., risk factors), prevention (e.g., safe sex and PrEP), and testing.
  Arms: Usual care group

SUMMARY:
HIV-serodiscordant male couples, in which one male partner is HIV-seropositive and the other is HIV-seronegative, experience multiple risks in HIV care and prevention. As stigma often hinders such couples' access to support and services, leveraging their relational resources is crucial for optimizing their outcomes. The proposed study will assess the efficacy of the three-session We-INtervention focusing on their relationship dynamics to enhance Chinese HIV-serodiscordant male couples' health and well-being.

A total of 160 Chinese HIV-serodiscordant male couples (320 individuals: 160 HIV-seropositive and 160 HIV-seronegative) will be randomized at a 1:1 ratio to either the intervention or control arm. In the intervention arm, the We-INtervention will be delivered to both partners of each couple separately. In the control arm, each couple will receive health information pamphlets.

DETAILED DESCRIPTION:
A pilot randomized controlled trial has already demonstrated the feasibility, acceptability, cultural sensitivity, and preliminary efficacy of the We-INtervention in improving the quality of life, psychological well-being, relationship satisfaction, and health behaviors of both partners in HIV-serodiscordant male couples. The proposed randomized controlled trial will extend the pilot study to examine the effects of the We-INtervention on stigma perception and other HIV-related behavioral outcomes, the mediators that account for the intervention effects, and the conditions under which the intervention is most effective.

The We-INtervention, if found to be effective, will be a valuable supplement to existing medical care modules.

ELIGIBILITY:
Inclusion criteria:

1. both partners are male,
2. both partners are aged 18 or above,
3. both partners report being in a committed relationship for at least 3 months,
4. one partner is HIV-seropositive and the other partner is HIV-seronegative (i.e., serodiscordant couple),
5. both partners have disclosed their serostatus to each other, and
6. both partners are willing to participate in this study.

Exclusion criteria:

1. either partner is unable to complete the assessment due to a low education level or to physical or psychological constraints and
2. either partner has been diagnosed with another chronic disease (e.g., cancer and coronary heart disease).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only male couples will be recruited.
Enrollment: 320 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Stigma | pre-intervention, post-intervention (upon the completion of intervention), 1-month follow-up, and 3-month follow-up.
  Stigma related to HIV status and homosexual identity will be assessed using the modified version of Negative Self-image Subscale of Berger's HIV Stigma Scale (Berger, Ferrans, & Lashley, 2001) with parallel items related to "being HIV seropositive" (HIV-seronegative partners will respond to "being a partner to someone who is HIV seropositive") and "being homosexual." This dual stigma assessment was used in the PI's previous study (Chen et al., 2020). Possible scores range from 0 (no stigma) to 39 (most stigma).
Quality of life (WHOQol-HIV for seropositive partners and WHOQol for seronegative partners) | pre-intervention, post-intervention (upon the completion of intervention), 1-month follow-up, and 3-month follow-up.
  Quality of life will be measured using the 29-item World Health Organization Quality of Life-HIV for the HIV-seropositive partners and the 24-item World Health Organization Quality of Life for the HIV-seronegative partners (WHO, 1998). These two measures were previously used in the PI's study of Chinese HIV-serodiscordant couples (Hou et al., 2023). Possible scores range from 0 (worst quality of life) to 108 (Best quality of life) for HIV-seropositive partners , and from 0 (worst quality of life) to 96 (Best quality of life) for HIV-seronegative partners.
Psychological well-being | pre-intervention, post-intervention (upon the completion of intervention), 1-month follow-up, and 3-month follow-up.
  Psychological well-being will be measured using the five-item WHO Well-Being Index (Topp et al., 2015). This scale was used in the PI's study of Chinese HIV-seropositive partners (Huang et al., 2018). Both partners will answer this scale. Items are scored on a six-point scale (0-5). The total score for this scale is calculated by summing all items. The score range is 0-25. Higher scores indicate a higher level of well-being.
Sexual behavior | pre-intervention, post-intervention (upon the completion of intervention), 1-month follow-up, and 3-month follow-up.
  Sexual behavior will be assessed via the participants' self-reports of condomless sex with their primary partner or any outside partner and of their partners' HIV status. Sexual agreement on the monogamous relationship will also be assessed. These items were previously used in Dr. Darbes's couple-focused interventions (e.g., Gamarel et al., 2020).
HIV-seropositive partners' ART adherence | pre-intervention, post-intervention (upon the completion of intervention), 1-month follow-up, and 3-month follow-up.
  HIV-seropositive partners' ART adherence will be measured using a visual analog scale to indicate missing doses (Zhang et al., 2020), previously used by the PI in an HIV-related RCT (GRF 11606221). Possible scores range from 0 (never adhere) to 10 (always adhere); and (b) single-item questions asking about missing and delayed doses in the last three days, seven days (one week) and 30 days (one month).
HIV-seronegative partners' PrEP use | pre-intervention, post-intervention (upon the completion of intervention), 1-month follow-up, and 3-month follow-up.
  HIV-seronegative partners' PrEP use will assess their knowledge of PrEP, their lifetime and current use of PrEP, and their willingness to use PrEP in their current relationship. These items were previously used in Dr. Darbes's couple-focused interventions (e.g., Gamarel et al., 2020). Self-report history of any lifetime PrEP use (yes/no), reason for taking PrEP (if relevant), PrEP use during the past month (yes/no), current PrEP use (yes/no), reasons for PrEP discontinuation (if relevant), number of PrEP pills taken every week during the past month (if relevant), frequency of missing PrEP pills during the past month (if relevant; 0=never to 3=often), strategic PrEP dosing (yes/no), type of strategic dosing schedule (if relevant), date of last dose of PrEP.

SECONDARY OUTCOMES:
We-disease appraisal | pre-intervention, post-intervention (upon the completion of intervention), 1-month follow-up, and 3-month follow-up.
  We-disease appraisal will be measured to assess the couples' appraisals of HIV ownership using modified items of the Inclusion of Other in the Self Scale (Aron et al., 1992). The PI previously used these modified items for research on Chinese HIV-serodiscordant couples (Hou et al., 2023). Both partners will answer this scale. The total score is based on this single item. The score range is 0-6. Higher scores indicate a higher level of we-disease appraisal.
Communication | pre-intervention, post-intervention (upon the completion of intervention), 1-month follow-up, and 3-month follow-up.
  Communication will be measured to assess how the couples handle arguments and communicate about disagreements using 16 items. This measurement was previously conducted by Dr. Darbes in a recent couple-focused intervention (Gamarel et al., 2020) and will be validated for the proposed study.Possible scores range from 0 to 64, with a higher score indicating a higher level of communication.
Common dyadic coping | pre-intervention, post-intervention (upon the completion of intervention), 1-month follow-up, and 3-month follow-up.
  Common dyadic coping will be assessed using the five-item subscale for common dyadic coping (e.g., coping with the problem together) of the Dyadic Coping Inventory (Bodenmann, 2008). The PI previously used it for research on Chinese HIV-serodiscordant couples (Hou et al., 2023). The total score for this scale is calculated by summing all items. The score range is 0-20. Higher scores indicate a higher level of common dyadic coping.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Fangzhouai Garden, Xiamen, Fujian
  - Guangzhou Yuele Healthcare Service Center, Guangzhou, Guangdong
  - Community Always There, Shenzhen, Guangdong
  - Jin Tang Six-Color Rainbow Healthcare Center, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shiu CS, Chen WT, Simoni J, Fredriksen-Goldsen K, Zhang F, Zhou H. The Chinese Life-Steps Program: A Cultural Adaptation of a Cognitive-Behavioral Intervention to Enhance HIV Medication Adherence. Cogn Behav Pract. 2013 May;20(2):202-212. doi: 10.1016/j.cbpra.2012.05.005. PMID 23667305
- [Result] Pan S, Sun S, Li X, Chen J, Xiong Y, He Y, Pachankis JE. A pilot cultural adaptation of LGB-affirmative CBT for young Chinese sexual minority men's mental and sexual health. Psychotherapy (Chic). 2021 Mar;58(1):12-24. doi: 10.1037/pst0000318. Epub 2020 Jun 15. PMID 32538644
- [Result] Gamarel KE, Sevelius JM, Neilands TB, Kaplan RL, Johnson MO, Nemoto T, Darbes LA, Operario D. Couples-based approach to HIV prevention for transgender women and their partners: study protocol for a randomised controlled trial testing the efficacy of the 'It Takes Two' intervention. BMJ Open. 2020 Oct 15;10(10):e038723. doi: 10.1136/bmjopen-2020-038723. PMID 33060086
- [Result] Burton J, Darbes LA, Operario D. Couples-focused behavioral interventions for prevention of HIV: systematic review of the state of evidence. AIDS Behav. 2010 Feb;14(1):1-10. doi: 10.1007/s10461-008-9471-4. PMID 18843530